CLINICAL TRIAL: NCT05905432
Title: A Randomized Double-blinded Phase 1 Clinical Trial to Assess Safety, Tolerability and Reactogenicity of the Pan-Malaria Transmission-Blocking Vaccine AnAPN1 in Healthy Adults Living in Gabon
Brief Title: Pan-Malaria Transmission-Blocking Vaccine AnAPN1
Acronym: PamTBVac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Global Health Innovative Technology Fund (Other)
Responsible Party: Principal Investigator, Prof. Ayola Akim ADEGNIKA, Professor, Centre de Recherche Médicale de Lambaréné
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AnAPN1
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Malaria
Keywords: transmission blocking
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dosage A1 (Experimental): n=2 will receive a dose of 20 mcg UF6b (A1), n=9 will receive 20 mcg AnAPN1: GLA-LSQ (5 mcg GLA/2 mcg LSQ) (A2)
  Interventions: Drug: Vaccine AnAPN1
- Dosage B1 (Experimental): n=2 will receive 50 mcg UF6b (B1), n=9 will receive 50 mcg UF6b: GLA- LSQ (12.5 mcg GLA/5 mcg LSQ) (B2)
  Interventions: Drug: Vaccine AnAPN1
- Dosage C1 (Experimental): n=2 will receive 100 mcg UF6b (C1); n=9 will receive 100 mcg UF6b: GLA- LSQ (25 mcg GLA/10 mcg LSQ) (C2)
  Interventions: Drug: Vaccine AnAPN1

INTERVENTIONS:
Drug: Vaccine AnAPN1 — AnAPN1 is a recombinant protein expressed in Escherichia coli. It consists of the UF6b construct, derived from the sequence of the Anopheles gambiae alanyl aminopeptidase N (XM_318000.4) and will be formulated with or without Synthetic Glucopyranosyl Lipid A (GLA)- LSQ adjuvant. Route of administration is intramuscular.

SUMMARY:
Malaria is still responsible for more than 627,000 deaths each year, predominantly among children under 5 years old. Current reductions in deaths have stagnated, and additional setbacks for malaria control programs due to the Coronavirus Disease 2019 (COVID-19) pandemic are expected. To achieve malaria elimination and eradication a leverage concerted approaches to reduce clinical disease and prevent new infections is a must. The existing malaria controls tools including the a recombinant protein-based malaria vaccine (RTS,S ,(trade name MosquirixMosquirix )), a malaria vaccine currently undergoing implementation studies and endorsed by the World Health Organization on October 7, 2021, can reduce disease burden for patients but cannot ultimately support malaria elimination and eradication since their effect on malaria transmission is at most partial. Consequently, complementary interventions, such as transmission-blocking vaccines (TBVs) may prove to be a cost-effective intervention that can reduce on-going residual transmission and the cascade of new infections.

DETAILED DESCRIPTION:
TBVs work by blocking parasite transmission to and from mosquitoes, with the added benefit of preventing the spread of parasites that have developed drug resistance or those that are vaccine-escape mutants of e.g. RTS,S. However, blocking transmission of all malaria species will be mandatory to achieve a globally relevant impact on malaria morbidity and mortality with Plasmodium falciparum and Plasmodium vivax being the most relevant targets. To date, the mosquito recombinant protein antigen vaccine Anopheline Alanyl Aminopeptidase N (AnAPN1)is the only TBV candidate that meets this need, wherein antibodies to this vaccine block both human malaria parasite species, underscoring its potential for supporting malaria elimination. The AnAPN1 vaccine consists of the AnAPN1 dimer antigen construct (UF6b) construct derived from the sequence of a protein of the mosquito midgut (Anopheles gambiae alanyl aminopeptidase), expressed as a recombinant protein in bacteria. With Global Health Innovative Technology Fund( GHIT) (G2020-208) support, the AnAPN1 reaches the First-In-Human milestone.

ELIGIBILITY:
Inclusion Criteria :

* Healthy male and female volunteers aged 18-45 years.
* Able and willing (in the investigator's opinion) to comply with all trial requirements.
* General good health based on medical history and clinical examination.
* Written informed consent.
* Available to participate in follow up for the duration of trial (6 months following the last injection).
* Reachable by phone during the whole trial period.
* Women only: Must agree to practice continuous effective contraception for the duration of the trial.

Exclusion Criteria:

* Positive for P. falciparum sexual and asexual stages by thick blood smear microscopy on admission and documented parasitologically confirmed malaria parasites of at least 1000 parasite/microliter in the past four weeks.
* Pregnancy, lactation, or intention to become pregnant during the trial.
* Previous participation in a malaria vaccine trial.
* HIV and microscopically detectable schistosomiasis and Soil-Transmitted helminth infection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Adverse events related to the vaccination. | Day 14
  Number and grade of adverse events possibly, likely, and definitely related to vaccination.

SECONDARY OUTCOMES:
anti-UF6b IgG concentration | Day 28
  Area under the curve of anti-UF6b immunoglobulin G (IgG) concentration, using a qualified and validated ELISA protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ayôla Akim ADEGNIKA, Principal Investigator — Centre de Recherches Medicales de Lambarene; Rhoel DINGLASAN, Study Director — University of Florida
Locations (1):
- Centre de Recherches Médicales de Lammbaréné, Lambaréné, Moyen-Ogooué Province, Gabon

IPD SHARING:
Plan to Share IPD: No